CLINICAL TRIAL: NCT01948739
Title: NRI:BMI Control of a Therapeutic Exoskeleton
Brief Title: Brain Machine Interface Control of an Robotic Exoskeleton in Training Upper Extremity Functions in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: University of Houston (Other); The Methodist Hospital Research Institute (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); TIRR Memorial Hermann (Other)
Responsible Party: Principal Investigator, Marcia k. O'Malley, Associate Professor of Mechanical Engineering, William Marsh Rice University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-13-0054; 1R01NS081854 (NIH)
Record Dates: First submitted 2013-06-21; First posted 2013-09-24 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Stroke; Hemiparesis
Keywords: Brain machine interface; Rehabilitation robotics; Stroke; Hemiparesis
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- BMI control of MAHI Exo-II (Experimental): MAHI EXO-II exoskeleton augmented with BMI system will be used to actively include the patient in the control loop, thereby making the therapy 'active' and engaging patients with various impairment severity in rehabilitation tasks. Patients will receive longitudinal training with the BMI-robotic interface for 3-4 sessions per week, over a period of 3 months.
  Interventions: Device: MAHI EXO-II exoskeleton augmented with BMI system

INTERVENTIONS:
Device: MAHI EXO-II exoskeleton augmented with BMI system — In this longitudinal study, adult subjects with hemiparesis due to acute or chronic stroke will receive robotic-assisted training through an EEG-based BMI control of robotic exoskeleton to study the changes in upper extremity motor function, cortical plasticity (using the EEG and fMRI). The training will be provided 3x/week for 12 sessions over one-month period.
  Other Names: Brain Machine Interface System; Rehabilitation robotics

SUMMARY:
The purpose of this study is:

1. To augment the MAHI Exo-II, a physical human exoskeleton, with a non-invasive brain machine interface (BMI) to actively include patient in the control loop and thereby making the therapy 'active'.
2. To determine appropriate robotic (kinematic data acquired through sensors on robotic device ) and electrophysiological ( electroencephalography- EEG based) measures of arm motor impairment and recovery after stroke.
3. To demonstrate that the BMI controlled MAHI Exo-II robotic arm training is feasible and effective in improving arm motor functions in sub-acute and chronic stroke population.

DETAILED DESCRIPTION:
This study aims to provide an adjunct to accelerate neurorehabilitation for stroke patients. The MAHI EXO-II, a physical human-robot interface, will be combined with a non-invasive brain-machine interface (BMI) to actively include the patient in the training of upper extremity motor functions.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of unilateral cortical and subcortical stroke confirmed by brain CT or MRI scan;
2. Subacute or chronic stroke; interval of at least 3month and interval of at least 6 months from stroke to time of enrollment, respectively;
3. No previous clinically defined stroke;
4. Age between 18-75 years;
5. Upper-extremity hemiparesis associated with stroke (manual muscle testing score of at least 2, but no more than 4/5 in the elbow and wrist flexors);
6. No joint contracture or severe spasticity in the affected upper extremity: i.e., significant increase in muscle tone against passive ROM is no more than ½ of full range for given joint e.g., elbow, wrist and forearm movements.
7. Sitting balance sufficient to participate with robotic activities;
8. No neglect that would preclude participation in the therapy protocol;
9. Upper limb proprioception present ( as tested by joint position sense of wrist);
10. No history of neurolytic procedure to the affected limb in the past four months and no planned alteration in upper-extremity therapy or medication for muscle tone during the course of the study;
11. No medical or surgical condition that will preclude participation in an occupational therapy program, that includes among others, strengthening, motor control and functional re-training of the upper limbs;
12. No contraindication to MRI;
13. No condition (e.g., severe arthritis, central pain) that would interfere with valid administration of the motor function tests;
14. English-language comprehension and cognitive ability sufficient to give informed consent and to cooperate with the intervention.-

Exclusion Criteria:

1. Orthopedic limitations of either upper extremity that would affect performance on the study;
2. Untreated depression that may affect motivation to participate in the study;
3. Subjects who cannot provide self-transportation to the study location.

Inclusion and Exclusion Criteria for Health Subjects:

Inclusion criteria:

* able to understand and sign the consent form
* age 18-65

Exclusion criteria: - Previous history of or MRI findings consistent with brain tumors, strokes, trauma or arterial venous malformations - Contraindication to MRI - Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-09-24 (Actual); Primary Completion 2018-04-28 (Actual); Study Completion 2018-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia K. O'Malley, PhD, Principal Investigator — William Marsh Rice University; Jose L. Contreras-Vidal, PhD, Principal Investigator — University of Houston; Gerard Francisco, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Robert G. Grossman, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- The Institute for Rehabilitation and Research (TIRR) at Memorial Hermann, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] A. Gupta, V. Patolgu, M.K. O'Malley, and C.M. Burgar (2008). Design, Control and Performance of RiceWrist: A Force Feedback Wrist Exoskeleton for Rehabilitation and Training, International Journal of Robotics Research (IJRR) 27(2): 233-51.
- [Background] Bradberry TJ, Gentili RJ, Contreras-Vidal JL. Fast attainment of computer cursor control with noninvasively acquired brain signals. J Neural Eng. 2011 Jun;8(3):036010. doi: 10.1088/1741-2560/8/3/036010. Epub 2011 Apr 15. PMID 21493978
- [Background] Yozbatiran N, Berliner J, O'Malley MK, Pehlivan AU, Kadivar Z, Boake C, Francisco GE. Robotic training and clinical assessment of upper extremity movements after spinal cord injury: a single case report. J Rehabil Med. 2012 Feb;44(2):186-8. doi: 10.2340/16501977-0924. PMID 22334347
- [Background] Bhagat NA, French J, Venkatakrishnan A, Yozbatiran N, Francisco GE, O'Malley MK, Contreras-Vidal JL. Detecting movement intent from scalp EEG in a novel upper limb robotic rehabilitation system for stroke. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:4127-4130. doi: 10.1109/EMBC.2014.6944532. PMID 25570900
- [Background] Bhagat NA, Venkatakrishnan A, Abibullaev B, Artz EJ, Yozbatiran N, Blank AA, French J, Karmonik C, Grossman RG, O'Malley MK, Francisco GE, Contreras-Vidal JL. Design and Optimization of an EEG-Based Brain Machine Interface (BMI) to an Upper-Limb Exoskeleton for Stroke Survivors. Front Neurosci. 2016 Mar 31;10:122. doi: 10.3389/fnins.2016.00122. eCollection 2016. PMID 27065787
- [Result] Bhagat NA, Yozbatiran N, Sullivan JL, Paranjape R, Losey C, Hernandez Z, Keser Z, Grossman R, Francisco GE, O'Malley MK, Contreras-Vidal JL. Neural activity modulations and motor recovery following brain-exoskeleton interface mediated stroke rehabilitation. Neuroimage Clin. 2020;28:102502. doi: 10.1016/j.nicl.2020.102502. Epub 2020 Nov 19. PMID 33395991
- See also: Mechatronics and Haptic Interfaces (MAHI) Lab (Dr.O'Malley, Rice Uni) — http://mahilab.rice.edu/
- See also: University of Houston Brain-Machine Interface System Team (Dr.Contreras-Vidal, UH) — http://www.facebook.com/UHBMIST
- See also: The UTHealth Motor Recovery Lab at TIRR Memorial Hermann Hospital (Dr.Francisco, UTHealth) — https://med.uth.edu/pmr/research/neuromodulation-and-neural-interfaces-research/
- Available data/document: Study Protocol — https://www.ncbi.nlm.nih.gov/pubmed/25570900

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 18 were enrolled and allocated to the intervention, but only 10 received the intervention.
Period: Overall Study
Arm/Group | BMI Control of MAHI Exo-II
Started | 18
Received Intervention | 10
Completed | 10
Not Completed | 8

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for those who received the intervention.
Arm/Group | BMI Control of MAHI Exo-II
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  Black or African American | 2
  Hispanic | 2
  White | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Stroke Type [Count of Participants; unit: Participants]
  Hemorrhagic stroke | 5
  Ischemic stroke | 5
Stroke Location [Count of Participants; unit: Participants]
  Cortical lesion | 4
  Subcortical lesion | 4
  Cortical and subcortical lesion | 2
Months Since Stroke [Mean (Standard Deviation); unit: months] | 37.4 (34.0)
Paretic Arm [Count of Participants; unit: Participants]
  Right | 5
  Left | 5
Fugl-Meyer Assessment-Upper Extremity (FMA-UE) [Mean (Standard Deviation); unit: score on a scale] — FMA is a stroke-specific, performance based impairment index. It quantitatively measures impairment based on Twitchell and Brunnstrom's concept of sequential stages of motor return in hemiplegic stroke patients. It uses an ordinal scale for scoring of 33 items for the upper limb component of the F-M scale (0:can not perform; 1:can perform partially; 2:can perform fully). Total range is 0-66, 0 being poor and 66 normal.
  score on a scale | 37.8 (11.7)
Action Research Arm Test (ARAT) [Mean (Standard Deviation); unit: score on a scale] — The ARAT is used to assess subject's ability to manipulate-lift-release objects horizontally and vertically, which differs in size, weight and shape. The test consists of 19 items divided into 4 sub-tests (grasp, grip, pinch, gross arm movement) and each item is rated on a 4-point scale. The possible total score ranges between 0-57. Higher scores indicate better performance.
  score on a scale | 25.3 (16.8)
Jebsen-Taylor Hand Function Test (JTHFT) [Mean (Standard Deviation); unit: items completed per second] — The JTHFT is a motor performance test and assesses the time needed to perform 7 everyday activities (for example, flipping cards and feeding). Score is reported as completed items per second.
  items completed per second | 1.046 (0.930)
NIH Stroke Scale (NIHSS) [Mean (Standard Deviation); unit: score on a scale] — The levels of stroke severity as measured by the NIHSS scoring system are: 0 = no stroke. 1-4 = minor stroke. 5-15 = moderate stroke. 15-20 = moderate/severe stroke.
  score on a scale | 3.4 (1.4)
Grip Strength [Mean (Standard Deviation); unit: kilograms of force] — A grip dynamometer will be used to measure maximum gross grasp force.
  kilograms of force | 11.13 (8.7)
Pinch Strength [Mean (Standard Deviation); unit: kilograms of force] — A pinch gauge will be used to measure maximum pinch force.
  kilograms of force | 4.48 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fugl-Meyer Arm (FMA) Motor Score
Description: FMA is a stroke-specific, performance based impairment index. It quantitatively measures impairment based on Twitchell and Brunnstrom's concept of sequential stages of motor return in hemiplegic stroke patients. It uses an ordinal scale for scoring of 33 items for the upper limb component of the F-M scale (0:can not perform; 1:can perform partially; 2:can perform fully). Total range is 0-66, 0 being poor and 66 normal.
Time Frame: Baseline, immediately after end of treatment (within a week), 2 weeks after end of treatment, 12 weeks after end of treatment
Population: 2 weeks after end of treatment, data for this outcome measure were not collected for 3 participants. 12 weeks after end of treatment, data for this outcome measure was not collected for 1 participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BMI Control of MAHI Exo-II
Number analyzed (Participants) | 10
score on a scale
  Baseline | 37.8 (11.7)
  Immediately after end of treatment (within a week) | 41.3 (11.9)
  2 weeks after end of treatment: number analyzed (Participants) | 7
  2 weeks after end of treatment | 47 (10.5)
  12 weeks after end of treatment: number analyzed (Participants) | 9
  12 weeks after end of treatment | 41.3 (12.9)

2. Primary Outcome: Neural Activity (Cortical Dynamics) Measured by Electroencephalography (EEG) Movement-related Cortical Potential (MRCP) Amplitude
Description: EEG activity in the low-frequency delta band will be assessed. Scalp EEG electrodes will be located over the motor cortex, specifically, central (Cz, C1- C4), fronto- central (FCz, FC1 - FC4) and centro-parietal electrodes (CPz, CP1 - CP4). Further, to account for left hand vs. right hand impairment, the electrode locations will be flipped for individuals with right hand impairment. Increased MRCP amplitude indicates increased activation of the ipsi-lesional hemisphere or inhibition of competing contra-lesional hemisphere, following motor relearning.
Time Frame: Baseline, immediately after end of treatment (within a week)
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | BMI Control of MAHI Exo-II
Number analyzed (Participants) | 10
microvolts
  Baseline | -1.49 (1.61)
  Immediately after end of treatment (within a week) | -1.66 (1.53)

3. Primary Outcome: Cortical Dynamics Measured by Electroencephalography (EEG) Movement-related Cortical Potential (MRCP) Latency
Description: EEG activity in the low-frequency delta band will be assessed. Scalp EEG electrodes will be located over the motor cortex, specifically, central (Cz, C1- C4), fronto- central (FCz, FC1 - FC4) and centro-parietal electrodes (CPz, CP1 - CP4). Further, to account for left hand vs. right hand impairment, the electrode locations will be flipped for individuals with right hand impairment. MRCP latency is the duration of MRCP prior to movement onset, and is defined as time difference starting from 50% of peak amplitude until the time of movement onset. Increased MRCP latency indicates increased activation of the ipsi-lesional hemisphere or inhibition of competing contra-lesional hemisphere, following motor relearning.
Time Frame: Baseline, immediately after end of treatment (within a week)
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | BMI Control of MAHI Exo-II
Number analyzed (Participants) | 10
milliseconds
  Baseline | 486.10 (92.56)
  Immediately after end of treatment (within a week) | 459.90 (109.60)

4. Primary Outcome: Movement Quality as Assessed by Exoskeleton Kinematics - Average Speed
Description: A higher value indicates better movement quality.
Time Frame: Baseline, immediately after end of treatment (within a week)
Measure: Mean (Standard Deviation); unit: degrees per second
Arm/Group | BMI Control of MAHI Exo-II
Number analyzed (Participants) | 10
degrees per second
  Baseline | 15.80 (8.28)
  Immediately after end of treatment (within a week) | 20.08 (7.29)

5. Primary Outcome: Movement Quality as Assessed by Exoskeleton Kinematics - Spectral Arc Length
Description: Spectral Arc Length is a frequency-domain measure that increases in value as movements become less jerky. A higher value indicates better movement quality (that is, movements are less jerky).
Time Frame: Baseline, immediately after end of treatment (within a week)
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | BMI Control of MAHI Exo-II
Number analyzed (Participants) | 10
unitless
  Baseline | -2.64 (0.95)
  Immediately after end of treatment (within a week) | -2.29 (0.47)

6. Primary Outcome: Movement Quality as Assessed by Exoskeleton Kinematics - Number of Peaks
Description: Number of peaks is a metric related to the shape of the velocity profile. A higher number of peaks implies jerkier movement. A lower number of peaks indicates better movement quality (that is, movements are less jerky).
Time Frame: Baseline, immediately after end of treatment (within a week)
Measure: Mean (Standard Deviation); unit: number of peaks
Arm/Group | BMI Control of MAHI Exo-II
Number analyzed (Participants) | 10
number of peaks
  Baseline | 2.13 (0.76)
  Immediately after end of treatment (within a week) | 1.78 (0.81)

7. Primary Outcome: Movement Quality as Assessed by Exoskeleton Kinematics - Time to First Peak
Description: Time to 1st Peak is a metric related to the shape of the velocity profile, and is reported as [(time to first peak) divided by (total movement duration)]. This value is usually less than the ideal value of 0.5, or 50%, of the total movement duration when a movement has more than one peak. The closer the value is to the ideal value of 0.5, the more well-balanced are the movements.
Time Frame: Baseline, immediately after end of treatment (within a week)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BMI Control of MAHI Exo-II
Number analyzed (Participants) | 10
seconds
  Baseline | 0.35 (0.14)
  Immediately after end of treatment (within a week) | 0.43 (0.16)

8. Secondary Outcome: Score on Action Research Arm Test (ARAT)
Description: The ARAT is used to assess subject's ability to manipulate-lift-release objects horizontally and vertically, which differs in size, weight and shape. The test consists of 19 items divided into 4 sub-tests (grasp, grip, pinch, gross arm movement) and each item is rated on a 4-point scale. The possible total score ranges between 0-57. Higher scores indicate better performance.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BMI Control of MAHI Exo-II
Number analyzed (Participants) | 10
score on a scale
  Baseline | 25.30 (16.80)
  Immediately after end of treatment (within a week) | 30.50 (20.89)
  2 weeks after end of treatmen | 34.71 (17.16)
  12 weeks after end of treatment | 30.33 (21.49)

9. Secondary Outcome: Score on Jebsen-Taylor Hand Function Test (JTHFT)
Description: The JTHFT is a motor performance test and assesses the time needed to perform 7 everyday activities (for example, flipping cards and feeding). Score is reported as items completed per second.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: activities completed per second
Arm/Group | BMI Control of MAHI Exo-II
Number analyzed (Participants) | 10
activities completed per second
  Baseline | 1.05 (0.93)
  Immediately after end of treatment (within a week) | 1.00 (0.88)
  2 weeks after end of treatment | 1.32 (0.86)
  12 weeks after end of treatment | 1.11 (0.88)

10. Secondary Outcome: Grip Strength
Description: A grip dynamometer will be used to measure maximum gross grasp force.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg of force
Arm/Group | BMI Control of MAHI Exo-II
Number analyzed (Participants) | 10
kg of force
  Baseline | 11.13 (8.70)
  Immediately after end of treatment (within a week) | 12.64 (9.91)
  2 weeks after end of treatment: number analyzed (Participants) | 7
  2 weeks after end of treatment | 13.33 (9.19)
  12 weeks after end of treatment: number analyzed (Participants) | 9
  12 weeks after end of treatment | 12.26 (9.42)

11. Secondary Outcome: Pinch Strength
Description: A pinch gauge will be used to measure maximum pinch force.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg of force
Arm/Group | BMI Control of MAHI Exo-II
Number analyzed (Participants) | 10
kg of force
  Baseline | 4.48 (2.29)
  Immediately after end of treatment (within a week) | 5.01 (2.53)
  2 weeks after end of treatment: number analyzed (Participants) | 7
  2 weeks after end of treatment | 5.47 (1.30)
  12 weeks after end of treatment: number analyzed (Participants) | 9
  12 weeks after end of treatment | 4.55 (1.45)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | BMI Control of MAHI Exo-II
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Absence of control group, low sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT01948739/Prot_SAP_000.pdf